CLINICAL TRIAL: NCT05244187
Title: Prospective, Multi-Center, Randomized Study to Evaluate the OrthoCor Active System for Pain Relief
Brief Title: Study to Evaluate the OrthoCor Active System for Pain Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Caerus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCM-OAS-01
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: 1:1 assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- OrthoCor Active System (Experimental): OrthoCor Active System used for pain relief
  Interventions: Device: OrthoCor Active System
- Standard of care (No Intervention): standard of care: over-the-counter pain medication

INTERVENTIONS:
Device: OrthoCor Active System — The OrthoCor Active System is a portable (battery operated) non-invasive device that delivers Pulsed Electromagnetic Field (PEMF) therapy for General Use of temporary pain relief, utilizing wraps that position the therapy, such as on the ankle, back, knee, wrist, elbow, shoulder, foot, or neck.
  Arms: OrthoCor Active System

SUMMARY:
This is a prospective, multi-center, randomized, pivotal study to evaluate the OrthoCor Active System in individuals prescribed its use in comparison with the standard of care intervention for pain relief.

DETAILED DESCRIPTION:
According to the Centers for Disease Control and Prevention, 50 million adults in the United States have chronic daily pain, with 19.6 million adults experiencing high impact chronic pain that interferes with daily life or work activities. Clinical best practices may recommend a collaborative, multimodal, multidisciplinary, patient-centered approach to treatment for various acute and chronic pain conditions to achieve optimal patient outcomes. For improved functionality, activities of daily living, and quality of life, clinicians are encouraged to consider and prioritize, when clinically indicated, nonpharmacologic approaches to pain management.

An alternative treatment option can be the use of restorative therapies. Restorative therapies play a significant role in acute and chronic pain management, and positive clinical outcomes are more likely if restorative therapy is part of a multidisciplinary treatment plan following a comprehensive assessment.

The OrthoCor Active System uses specialized Pulsed Electromagnetic Field (PEMF) technology to relieve pain and reduce edema through safe, clinically proven therapy. PEMF is a low-level, time-varying electromagnetic field that penetrates superficial soft tissue, helping to accelerate the body's natural anti-inflammatory and recovery responses. Inside every OrthoCor Active System is proprietary electronic circuitry that delivers PEMF to the source of injuries. PEMF has been shown to stimulate reaction pathways that result in pain and inflammation reduction. OrthoCor's patented PEMF accelerates the binding of calcium (Ca2+) to calmodulin (CaM), the process responsible for the body's natural, antiinflammatory nitric oxide (NO) cascade. NO is a key element in the body's natural healing process. It is also a vasodilator, increasing blood and lymphatic flow. Additionally, NO down-regulates interleukin-1 beta (IL1β) and inducible nitric oxide synthase (iNOS), which leads to reduced cyclooxygenase-2 (COX-2) and prostaglandins - molecules responsible for causing inflammation and pain. Unlike other systemic COX-2 inhibitors such as nonsteroidal anti-inflammatory drugs (NSAIDs), OrthoCor's targeted PEMF signals stimulate localized reaction pathways, thereby reducing pain and inflammation without the risks and side effects associated with NSAIDs.

In previous clinical studies, OrthoCor Active System was clinically proven to reduce pain, swelling and provide lasting relief without the use of pain medications or invasive procedures. OrthoCor Medical Inc. conducted a prospective, double blind, placebo controlled, randomized pilot study (2014-2016), enrolling 80 patients with Kellgren-Lawrence knee arthritis who used the OrthoCor knee system, which showed a significant 60% reduction in the mean pain score within the first 3 days of use compared with the sham group 2. A preliminary study conducted by OrthoCor Medical Inc. in 33 patients suffering from knee osteoarthritis utilizing the OrthCor knee system, showed reduced pain and stiffness after 15 days of treatment with a 43% reduction in pain score and a 79% improvement in activity limitations, symptoms, emotions, and overall quality of life.

The OrthoCor Active System is a portable (battery operated) non-invasive shortwave diathermy medical device which applies electromagnetic energy at a radio frequency (RF) of 27.12 MHz for the treatment of pain in superficial soft tissue, such as in the ankle, back, knee, wrist, elbow, shoulder, foot, or neck. The OrthoCor Active System delivers the pulsed RF signal of 6.5+0.5 Ws/cm3 to the tissue target via the inductive coupling with an applicator coil. The system also uses disposable, single-use, air activated OrthoPods that provide heat for the temporary relief of minor muscular & joint aches & pains associated with overexertion, strains, sprains, and arthritis.

The objective of this study is to evaluate the OrthoCor Active System in individuals presenting with post-operative pain and edema in superficial soft tissue. The OrthoCor Active System will be compared to the SOC intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals presenting with pain in superficial soft tissue, such as ankle, back, knee, wrist, elbow, shoulder, foot, or neck pain, or minor muscular and joint aches and pains associated with over exertion, strains, sprains, or arthritis
2. Prescribed use of the OrthoCor Active System or Standard of Care (SOC) intervention
3. Willing and able to provide informed consent or obtain consent from legal authorized representative (LAR)

Exclusion Criteria:

1. Have a cardiac pacemaker, cardioverter defibrillator, neurostimulator, infusion pump or any active medical implant
2. Have an implanted metallic lead or any type of wire coil implant, or any implanted system that may contain lead
3. Who are or may be pregnant
4. Have an open wound at the area of application
5. Are not capable or fully aware to the sensation of heat
6. Have poor circulation or heart disease
7. Have diabetes
8. Under the age of 18 or individuals with open bone growth plates
9. Unable to provide consent or obtain consent from a LAR
10. Unwilling or unable to use the OrthoCor Active System or Standard of Care (SOC) intervention
11. Unwilling or unable to complete the daily pain assessment
12. Enrolled in a study to evaluate an investigational drug
13. Prisoner or under incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua G Hackel, MD, Principal Investigator — Andrews Research and Education Foundation
Locations (5):
- United States (5):
  - Andrews Research & Education Foundation, Gulf Breeze, Florida
  - GFC of Southeastern Michigan PC, Detroit, Michigan
  - Rothman Orthopedic Institute, Washington Township, New Jersey
  - Orlin & Cohen Orthopedic Group, Smithtown, New York
  - Spinal Pain and Rehabilitation Medicine, Yonkers, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hackel JG, Paci JM, Gupta S, Maravelas DA, North TJ, Paunescu A. Evaluating Noninvasive Pulsed Electromagnetic Field Therapy for Joint and Soft Tissue Pain Management: A Prospective, Multi-center, Randomized Clinical Trial. Pain Ther. 2025 Apr;14(2):723-735. doi: 10.1007/s40122-025-00711-z. Epub 2025 Feb 10. PMID 39928254

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OrthoCor Active System | Standard of Care
Started | 59 | 61
Completed | 48 | 43
Not Completed | 11 | 18

BASELINE CHARACTERISTICS:
Population: The numbers represent the ITT because the analyses for PP and ITT are very similar.
Groups:
- Total: Total of all reporting groups
Arm/Group | OrthoCor Active System | Standard of Care | Total
Number analyzed (Participants) | 59 | 61 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (16.3) | 56.5 (16.2) | 55.3 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 39 | 78
  Male | 20 | 22 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 18 | 19 | 37
  White | 31 | 39 | 70
  More than one race | 5 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59 | 61 | 120

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety EndPoint
Description: Number of participants with adverse events
Time Frame: after 2 weeks of use
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | OrthoCor Active System | Standard of Care
Number analyzed (Participants) | 59 | 61
Participants | 2 | 2

2. Primary Outcome: Primary Efficacy EndPoint
Description: Change from baseline of Mankoski pain scale between OrthoCor and standard of care. The Mankoski pain scale ranges from 0 representing no pain to 10 representing pain causing unconsciousness.
Time Frame: at baseline compared to during 2 weeks of use
Population: PP
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | OrthoCor Active System | Standard of Care
Number analyzed (Participants) | 48 | 43
score on a scale | -1.8 [-2.1 to -1.5] | -0.5 [-0.8 to -0.1]

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: FDA definitions of adverse events was used and all events experienced by the patients were reported adn evaluated by a safety officer
Arm/Group | OrthoCor Active System | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/61
Other Adverse Events (participants affected / at risk) | 2/59 | 2/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OrthoCor Active System (N=59) | Standard of Care (N=61)
shoulder pain (Surgical and medical procedures) | 0 (0) | 1 (1)
tingling (Surgical and medical procedures) | 1 (1) | 0 (0)
difficulty bending knee (Surgical and medical procedures) | 1 (1) | 0 (0)
sleepiness (Social circumstances) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT05244187/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT05244187/SAP_001.pdf